CLINICAL TRIAL: NCT01385774
Title: SUPERvised Exercise Therapy (SET) or Immediate Percutaneous Transluminal Angioplasty (PTA) for Intermittent Claudication (IC) in Patients With an Iliac Artery Obstruction: A Randomized Controlled Trial. SUPER Study
Brief Title: SUPER Study; SUPERvised Exercise or Angioplasty for Intermittent Claudication Due to an Iliac Artery Obstruction.
Acronym: SUPER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated after 240 patients because of slow accrual and lack of additional funding
Sponsor: M.J.W. Koelemaij (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, M.J.W. Koelemaij, Dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171102025;ZonMw; 09/285;METC AMC (Other: Protocol number; IRB AMC Amsterdam)
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Intermittent Claudication; Peripheral Arterial Disease
Keywords: Intermittent Claudication; Percutaneous Transluminal Angioplasty; Supervised Exercise Therapy; Peripheral Arterial Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Angioplasty; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group: Angioplasty (Active Comparator): Angioplasty with or without stent of the iliac artery
  Interventions: Procedure: Percutaneous Transluminal Angioplasty
- Control: Supervised Exercise Therapy (Active Comparator): Supervised exercise therapy by a physiotherapist
  Interventions: Other: Supervised Exercise Therapy

INTERVENTIONS:
Procedure: Percutaneous Transluminal Angioplasty — The Percutaneous Transluminal Angioplasty (PTA) procedure will be performed by an experienced interventional radiologist using a conventional guide wire and balloon catheter technique. A stent will be placed in cases in which the residual mean pressure gradient is greater than 10 mmHg across the treated site or when more than 30% stenosis after the procedure is detected. All PTA patients are encouraged perform at least three walking sessions every day.
  Other Names: Endovascular treatment
  Arms: Intervention group: Angioplasty
Other: Supervised Exercise Therapy — Supervised Exercise Therapy (SET) will take place in the hospital or community based according to the guidelines of the Dutch Society for Physiotherapists. The duration of the treatment will be at least 6 months and with a frequency of 2 times a week for at least 60 minutes and an intensity near maximum pain barrier (defined as pain of which it is not possible to be distracted). The frequency of the training will decrease after 3 months and the patients will receive homework, make a plan and keep a log of their exercise activities. Furthermore the program consists of walking pattern improvement and enhancement of endurance and strength. All SET patients are encouraged to perform at least three walking sessions every day on their own.
  Other Names: Conservative treatment
  Arms: Control: Supervised Exercise Therapy

SUMMARY:
The purpose of our study is to compare the clinical effectiveness and cost-effectiveness of two treatment strategies of Intermittent Claudication (IC) due to an iliac artery obstruction: to start with SUPERvised Exercise Therapy (SET) and deferred Percutaneous Transluminal Angioplasty (PTA) in case of SET failure, or immediate PTA.

It is our hypothesis that PTA as first line treatment is more effective than SET as first line treatment with regard to maximum walking distance, quality of life and costs after one year.

DETAILED DESCRIPTION:
Intermittent claudication (IC) is a manifestation of cardiovascular disease, reflected by a threefold increased risk in these patients of developing serious cardiovascular events. Treatment of patients with IC is aimed at secondary prevention of cardiovascular events by control of risk factors for atherosclerotic disease, and to improve walking distance and subsequently quality of life. Supervised Exercise Therapy (SET) and Percutaneous Transluminal Angioplasty (PTA) can effectively improve pain free walking distance, but the optimal choice of treatment, specifically in patients with an iliac artery stenosis or occlusion is unclear. PTA is attractive as initial therapy since PTA of the iliac arteries has an immediate effect and it is durable. There is a lack of evidence from randomized controlled trials (RCT) to define the optimal treatment strategy for patients with IC due to iliac artery lesions; first line treatment with SET and PTA in case of failure, or immediate iliac artery PTA.

Purpose:

To define the optimal treatment strategy of IC due to an iliac artery obstruction: To start with SET and deferred PTA in case of SET failure, or immediate PTA.

Design:

Multicenter randomized controlled trial.

Patients:

400 patients with IC due to an iliac artery stenosis or occlusion.

Interventions:

SET and PTA.

Outcomes:

Primary outcomes are quality of life (Qol) recorded with the disease specific VascuQol instrument and maximum walking distance on a standardized treadmill test with a speed of 3.2 km/h at 10% incline after 1 year.

Secondary outcomes are pain-free walking distance, generic Qol, functional status, complications, number of treatment failures and costs. Economic evaluation comprises a cost-effectiveness and cost-utility analysis from a societal perspective, with the costs per patient able to walk maximal, respectively the costs per Quality Adjusted Life-Year (QALY) as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Disabling claudication as defined by surgeon based on patient's history;
3. Ankle/Brachial Index (ABI) < 0.9 or drop in ABI > 0.15 after exercise test;
4. Hemodynamic stenosis of the common or external iliac artery on Color Duplex Scanning (CDS) (PSV ratio ≥ 2.5 or EDV ≥ 0.6 m/s) or on Magnetic Resonance Angiography (MRA) or Computed Tomography Angiography (CTA)(> 50% stenosis) or occlusion of the common or external iliac artery on CDS (PSV 0 m/s) or on MRA or CTA;
5. Iliac artery lesion and a concomitant stenosis in the superficial femoral artery defined as stenosis > 50% by CDS (PSV ratio ≥ 2.5 or EDV ≥ 0.6 m/s) or on MRA or CTA, or occlusion on CDS (PSV 0 m/s) or MRA or CTA;
6. Lesion classified A, B or C according to the TASC (TransAtlantic Inter-Society Consensus) classification of aortoiliac lesions;
7. Patient is able to walk at least 2 minutes on a treadmill at 3.2 km/h and 10% incline;
8. The Maximum Walking Distance on a treadmill < 300 meters.

Exclusion Criteria:

1. Life expectancy < 3 months;
2. Patient is unable to complete self-reported questionnaires (insufficiently reading or speaking the Dutch language, cognitive disorders, etc);
3. Patient is unable to give informed consent;
4. A documented contrast allergy;
5. Pregnancy;
6. Contra-indication for anticoagulant therapy;
7. Duration of current complaints < 3 months;
8. Occlusion of the common femoral artery at the affected side;
9. Patient participates in another study;
10. Heart failure or Angina Pectoris NYHA III or IV. (NYHA III: Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea; NYHA IV: Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased);
11. Patient previously received Supervised Exercise Therapy (SET) according to KNGF (Dutch Society for Physiotherapists) guidelines;
12. Renal insufficiency (serum creatinin > 150 micromol/l).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Disease specific Quality of Life | 12 months
  Disease specific Quality of life (Qol) recorded with the disease specific VascuQol instrument 1 year after intervention.
  The VascuQol will be completed at baseline and 1,6,12 months follow-up.
Maximum Walking Distance | 12 months
  Maximum walking distance on a standardized treadmill test with a speed of 3.2 km/h at 10% incline measured 1 year after intervention.
  The maximum walking distance will be assessed at baseline and 1,6,12 months follow-up.

SECONDARY OUTCOMES:
Painfree Walking Distance | 12 months
  Painfree walking distance on a standardized treadmill test with a speed of 3.2 km/h at 10% incline 1 year after intervention.
  The painfree walking distance will be assessed at baseline and 1,6,12 months follow-up.
Functional Status | 12 months
  Functional status assessed by the AMC Linear Disability Score (ALDS) 1 year after intervention.
  The ALDS will be completed at baseline and 1,6,12 months follow-up.
Generic Quality of Life | 12 months
  Generic quality of life (Qol) recorded with the Short Form 36 (SF-36) and EQ-5D (former EuroQoL).
  The SF-36 will be completed at baseline and 1,6,12 months follow-up. The EQ-5D will be completed at baseline, 1 week and 1,6,12 months follow-up.
Complications | During 12 months
  Complications related to both interventions during 12 months.
Treatment failures | During 12 months
  A treatment failure is defined as crossover to the other treatment arm.
Costs | During 12 months
  Costs during 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mark JW Koelemay, M.D., Ph.D, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jim A Reekers, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Dink A Legemate, M.D.,Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Shandra Bipat, Ph.D., Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (15):
- Netherlands (15):
  - Flevoziekenhuis, Almere Stad
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - VU Medical Center, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academic Medical Center, Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Ziekenhuis Rijnstate, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Deventer Ziekenhuis, Deventer
  - Kennemer Gasthuis, Haarlem
  - Tergooiziekenhuizen, Hilversum
  - Spaarne Ziekenhuis, Hoofddorp
  - St Antonius Ziekenhuis, Nieuwegein
  - UMC St. Radboud, Nijmegen
  - Waterland ziekenhuis, Purmerend

REFERENCES:
- [Derived] Frans FA, Zagers MB, Jens S, Bipat S, Reekers JA, Koelemay MJ. The relationship of walking distances estimated by the patient, on the corridor and on a treadmill, and the Walking Impairment Questionnaire in intermittent claudication. J Vasc Surg. 2013 Mar;57(3):720-727.e1. doi: 10.1016/j.jvs.2012.09.044. Epub 2013 Jan 11. PMID 23313183
- [Derived] Frans FA, Bipat S, Reekers JA, Legemate DA, Koelemay MJ; SUPER Study Collaborators. SUPERvised exercise therapy or immediate PTA for intermittent claudication in patients with an iliac artery obstruction--a multicentre randomised controlled trial; SUPER study design and rationale. Eur J Vasc Endovasc Surg. 2012 Apr;43(4):466-71. doi: 10.1016/j.ejvs.2012.01.014. Epub 2012 Feb 10. PMID 22326696